CLINICAL TRIAL: NCT04676386
Title: Biomarker Analysis in High PD-L1 Expressing NSCLC Patients Treated With PD-1/PD-L1 Based Therapy With or Without the Addition of Platinum Based Chemotherapy
Acronym: BEACON-LUNG
Status: Terminated | Type: Observational
Why Stopped: Recruitment futility
Sponsor: Addario Lung Cancer Medical Institute (Other)
Collaborators: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ALCMI-014
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: NSCLC Stage IV; NSCLC, Stage IIIC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A maximum of three blood draws will be performed over three years.
  Approximately 25 mLs venous blood will be collected into blood collection tubes provided in the study kit. Blood should be drawn at the time of other clinical laboratories whenever possible to prevent additional venipuncture or port access, otherwise, a study-specific blood draw may occur at the time of the standard of care office visit.
  Peripheral blood draws may occur on-site or via a remote phlebotomist dispatched by the enrolling institution. Sites may mail the blood draw kit to the subject prior to arrival of the remote phlebotomist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PD1/PD-L1: Standard of Care: PD1/PD-L1 monotherapy
  Interventions: Diagnostic Test: Primary Immune Response (PIR) test by Biodesix, Inc.
- PD1/PD-L1 + chemo: Standard of Care: Platinum doublet-based chemotherapy plus PD-1/PD-L1 combination
  Interventions: Diagnostic Test: Primary Immune Response (PIR) test by Biodesix, Inc.

INTERVENTIONS:
Diagnostic Test: Primary Immune Response (PIR) test by Biodesix, Inc. — Blood draw for biomarker assessment will be performed at these time-points: pretreatment, start of 3rd cycle and investigator assessed progression. The biomarker analysis will be performed retrospectively.

SUMMARY:
This Observational study will explore the utility of the Biodesix, Inc. "PIR" (primary immune response) test to predict outcomes in treatment-naïve advanced stage NSCLC with PD-L1 tumor proportion score (TPS) > 50% and ECOG performance status (PS) 0-2 NSCLC patients who are treated with PD-1/PD-L1 based therapy with or without the addition of platinum based chemotherapy.

DETAILED DESCRIPTION:
This is an observational, multicenter study designed to assess biomarkers (serum and plasma) as predictive of early progression in 390 treatment-naive patients with advanced stage non-small cell lung cancer (NSCLC) and PD-L1 TPS ≥50% treated with two standard of care (SOC) regimens, platinum based PD-1/PD-L1 regimen with monotherapy (single agent PD-1/PD-L1 therapy).

Prior to enrollment, tumor specimens will be tested for PD-L1 expression according to participating centers' standard operating procedures. Patients will be treated, according to physician choice, with platinum-based PD-1/PD-L1 regimen versus single agent PD-1/PD-L1 regimen. For each treatment cohort of 195 patients, enrollment will proceed in sub-cohorts to ensure a population with 20% ECOG PS2 patients and a total of 40 squamous cell carcinoma patients per treatment arm.

Patients will receive one of the following standard-of-care (SOC) treatment regimens at the discretion of the treating investigator:

* PD-1/PD-L1 therapy
* Platinum doublet-based chemotherapy plus PD-1/PD-L1 combination

Tumor assessment will follow RECIST v1.1.

Blood draw for biomarker assessment will be performed at these time-points: pretreatment, start of 3rd cycle and investigator assessed progression. The biomarker analysis will be performed retrospectively.

Remaining serum and plasma will be stored for subsequent exploratory studies and will be available to the investigators in the ALCMI network per ALCMI standard operating procedures.

Additionally, pathology reports including PD-L1 results and Next Generation Sequencing results, from any CLIA laboratory, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naïve for their stage IIIC/IV AJCC 8 non-small cell lung cancer with a tumor biopsy PD-L1 TPS > 50%
* Intent to treat with PD-1/PD-L1 or PD-1/PD-L1 plus pemetrexed/carboplatin or paclitaxel/nab-paclitaxel/carboplatin
* ECOG PS 0-2
* Ability to consent to participate in the study

Exclusion Criteria:

* Ability to understand the requirements of the protocol or to provide informed consent is impaired or is unwilling to comply with the protocol requirements

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be treatment-naïve advanced NSCLC patients with PD-L1 TPS ≥50% who will receive PD-1/PD-L1 or PD-1/PD-L1 plus pemetrexed/carboplatin or paclitaxel/nab-paclitaxel/carboplatin and are managed per treating physician's standard of care.
Sampling Method: Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Biomarker PIR evaluation | 3 years
  To collect biospecimens and evaluate candidate biomarkers of early progression on patients with >50% PD-L1 positive tumors treated with PD-1/PD-L1 monotherapy or PD-1/PD-L1/chemotherapy combination

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Addario Lung Cancer Medical Institute (ALCMI), San Carlos, California
  - Rush University Medical Center, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Undecided